CLINICAL TRIAL: NCT02742662
Title: Smart Technology for Weight Loss and Metabolic Health- A Randomized Controlled Trial
Brief Title: Smart Technology for Weight Loss and Metabolic Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Temple University (Other)
Collaborators: The Obesity Treatment Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 23217
Record Dates: First submitted 2016-04-07; First posted 2016-04-19 (Estimated); Last update posted 2018-02-15 (Actual); Status verified 2018-02

CONDITIONS: Obesity; Overweight; Prediabetes; Weight Loss; Lifestyle
Keywords: Obesity; Overweight; Prediabetes; Smartphone application; Technology; Weight Loss; Lifestyle Intervention
MeSH Terms: conditions — Obesity; Overweight; Prediabetic State; Weight Loss | interventions — Wearable Electronic Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Smart Technology Group (Experimental): The Smart Technology Group will receive a technology-based lifestyle intervention program which uses wearable technology, smartscales and smartphone applications to track and deliver feedback on caloric expenditure, physical activity, caloric intake and body weight. Participants will receive information through smartphone applications on strategies to make changes to their diet, physical activity, and weight-related behaviors along with standard 3 monthly in-person weight management visits.
  Interventions: Device: Wearable technology, smartscale; Behavioral: Smartphone applications; Behavioral: Standard Weight Management Visits
- Standard Weight Management Group (Other): The Standard Weight Management Group will receive 3 monthly in-person weight management visits during which they will receive standard of care lifestyle recommendations in accordance with the 2013 American Heart Association/American College of Cardiology/The Obesity Society Guideline.
  Interventions: Behavioral: Standard Weight Management Visits

INTERVENTIONS:
Device: Wearable technology, smartscale
  Arms: Smart Technology Group
Behavioral: Smartphone applications
  Arms: Smart Technology Group
Behavioral: Standard Weight Management Visits

SUMMARY:
The study will evaluate whether a technology-based lifestyle intervention program using primarily a smartphone platform is an acceptable and effective way for treating obesity. The goal of the program is to achieve weight loss and enhance the health of overweight or obese subjects by improving their diet and activity via smartphone applications as compared with conventional in-person weight management programs.

ELIGIBILITY:
Inclusion Criteria:

* Overweight or obese BMI 25-42 kg/m2
* Employed in sedentary occupations
* Own a personal smartphone with unlimited data plan or >4 GigaByte data
* Proficient with use of smartphone applications and technology with current daily usage
* Ability to engage in moderate intensity exercise
* Weight stability for the last 2 months
* Participants must be willing to comply with all study-related procedures

Exclusion Criteria:

* Current or planned pregnancy
* Cardiovascular, pulmonary, renal disease, joint disease
* Uncontrolled thyroid disease
* History of eating disorders, psychiatric disease
* History of substance abuse or dependence in the last 1 year
* Diabetes
* Shift work
* Previous weight loss surgery
* Use of weight loss drugs/diet/program in the last 6 weeks
* Inability to increase walking as a form of exercise and to engage in moderate intensity exercise
* Other conditions or medications that affect body weight/appetite/metabolism
* Serious or unstable medical or psychological conditions that would compromise the subject's safety for successful participation
* Incapable of adhering with an intensive lifestyle intervention using technology and smartphone applications

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2016-04; Primary Completion 2017-06 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Change in body weight in kg | 6 months

SECONDARY OUTCOMES:
Change from baseline blood pressure | 6 months
Change from baseline waist circumference | 6 months
Change from baseline insulin resistance by homeostasis model assessment (HOMA-IR) | 6 months
Change from baseline hemoglobin A1c | 6 months
Change from baseline plasma triglycerides | 6 months
Change from baseline body weight in kg | 3 months
Change from baseline body weight in kg | 12 months
Change from baseline blood pressure | 12 months
Change from baseline waist circumference | 12 months
Change in Quality of Life | 6 months after receiving the intervention
  SF36 Questionnaire in wait-listed control group after the intervention
Change in insulin resistance by homeostasis model assessment (HOMA-IR) | 12 months compared to baseline and 6 months after receiving the intervention
  Wait-listed control group
Change in hemoglobin A1c | 12 months compared to baseline and 6 months after receiving the intervention and from baseline
  Wait-listed control group
Change in plasma triglycerides | 12 months compared to baseline and 6 months after receiving the intervention
  Wait-listed control group

CONTACTS AND LOCATIONS:
Overall Officials: Cherie Vaz, MD Dipl ABOM, Principal Investigator — Temple University
Locations (1):
- Temple University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No